CLINICAL TRIAL: NCT04099888
Title: A Multi-Center Randomised Open-Label Phase 2 Study to Assess the Safety, Tolerability and Efficacy of Fimaporfin-Induced Photochemical Internalisation of Gemcitabine Complemented by Gemcitabine/Cisplatin Chemotherapy Versus Gemcitabine/Cisplatin Alone in Patients With Inoperable Cholangiocarcinoma
Brief Title: PCI Treatment/Gemcitabine & Chemotherapy vs Chemotherapy Alone in Patients With Inoperable Extrahepatic Bile Duct Cancer
Acronym: RELEASE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recent results from a Phase 3 study are expected to change the standard of care for patients with inoperable CCA, rendering the RELEASE study challenging to complete and potentially inadequate for NDA approval.
Sponsor: PCI Biotech AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCIA 203/18
Record Dates: First submitted 2019-07-26; First posted 2019-09-23 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-04

CONDITIONS: Cholangiocarcinoma
Keywords: Phase II; Safety; Tolerability; Efficacy; Amphinex-induced Photochemical Internalisation; PCI; Amphinex; Gemcitabine; Cisplatin; Inoperable; CCA; Cholangiocarcinoma; Bile duct cancer; Photodynamic therapy; Extrahepatic; Perihilar; Distal; Fimaporfin; Pivotal; RELEASE; PDT; FimaChem; Klatskin; First line treatment; Standard of care; SOC; Chemotherapy; Local treatment
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Gemcitabine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PCI treatment in conjunction with Standard of Care (SoC) (Experimental): Arm A: Fimaporfin-induced photochemical internalisation (PCI) of gemcitabine complemented by gemcitabine/cisplatin chemotherapy
  Interventions: Drug: Fimaporfin and Gemcitabine; Drug: Gemcitabine/Cisplatin chemotherapy
- Standard of Care (SoC) (Active Comparator): Arm B: Gemcitabine/cisplatin chemotherapy
  Interventions: Drug: Gemcitabine/Cisplatin chemotherapy

INTERVENTIONS:
Drug: Fimaporfin and Gemcitabine — PCI treatment consists of IV administration of Amphinex solution for injection (investigational product) at 0.22 mg/kg dose of fimaporfin, followed 4 days later by a standard dose of gemcitabine infusion (1000 mg/m²) and intraluminal laser light application. Up to 2 PCI treatments will be given.
  Other Names: PCI treatment
  Arms: PCI treatment in conjunction with Standard of Care (SoC)
Drug: Gemcitabine/Cisplatin chemotherapy — Up to 8 cycles of gemcitabine/cisplatin combination chemotherapy will be administered.
  Other Names: Standard of care (SoC)

SUMMARY:
This study will assess the safety and effectiveness of fimaporfin-induced photochemical internalisation (PCI) of gemcitabine complemented by systemic gemcitabine/cisplatin chemotherapy compared to gemcitabine/cisplatin alone, in patients with inoperable cholangiocarcinoma (CCA). Participants will be randomly assigned to one of the treatment groups and will receive study treatment for 6 months, followed by assessments every 3 months, as applicable.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is an uncommon adenocarcinoma arising from cells lining the bile ducts. Standard treatment options for CCA include surgery, radiotherapy and chemotherapy, dependent upon if the CCA is intra- or extra-hepatic. Surgical removal of the tumor is the only potential cure, and CCA is very resistant to standard pharmaceutical drug treatment, though chemotherapy has some effect. Current chemotherapy uses cisplatin plus gemcitabine. Photochemical internalisation (PCI) is a novel technology, where photochemical reactions are used to enhance the effect of drugs by increasing their ability cross cell membranes to interact with their intended target. This study will assess the safety and effectiveness of fimaporfin-induced PCI of gemcitabine complemented by systemic gemcitabine/cisplatin chemotherapy compared to gemcitabine/cisplatin alone, in patients with inoperable CCA.

NOTE: Participants are no longer being recruited to this study.

ELIGIBILITY:
Inclusion Criteria:

1. Each patient must provide signed and witnessed written informed consent and agree to comply with study protocol requirements.
2. Histopathologically/cytologically verified adenocarcinoma consistent with cholangiocarcinoma (CCA). Must have biliary lesion causing bile obstruction that requires stenting and is accessible for PCI light treatment (ie, extrahepatic CCA [perihilar or distal] only).
3. CCA must be considered inoperable with respect to radical resection.
4. At least 1 radiologically evaluable lesion (measurable and/or non-measurable) that can be assessed at baseline and is suitable for repeated radiological evaluation.
5. If metastatic, metastases must be limited tissues other than bone or the central nervous system.
6. Must have adequate biliary drainage (at least 50% of the liver volume or at least 2 sectors) with no evidence of active uncontrolled infection (patients on antibiotics are eligible).
7. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Estimated life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Patients who have previously received any anti-tumor (either local or systemic) treatment for CCA, except for previous treatment of up to 2 cycles of gemcitabine/cisplatin.
2. Patients with severe visceral disease other than CCA.
3. A history of frequently recurring septic biliary events.
4. Patients with porphyria or hypersensitivity to porphyrins.
5. Patients with a second primary cancer with a disease-free interval of <5 years. A second primary cancer that has been treated with intent to cure may be allowed after consultation with the study Medical Monitor. Adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, in-situ carcinoma of the uterine cervix, or prostate cancer that is controlled by hormone therapy (patients may continue hormone therapy while on study) are allowed.
6. Patients not able to undergo contrast-enhanced CT or MRI.
7. Patients currently participating in any other interventional clinical trial.
8. Planned surgery, endoscopic examination or dental treatment in the first 30 days after PCI treatment.
9. Co-existing ophthalmic disease likely to require slit-lamp examination within the first 90 days after PCI treatment.
10. Clinically significant and uncontrolled cardiac disease except for extra systoles or minor conduction abnormalities and controlled and well-treated chronic atrial fibrillation.
11. Known allergy or sensitivity to photosensitisers (active substance and/or any of the excipients); or chronic use of other photosensitising therapies; treatment with amiodarone during the last 12 months.
12. Known hypersensitivity to or contraindication to the use of gemcitabine (active substance and/or any of the excipients).
13. Known hypersensitivity to or contraindication to the use of cisplatin (active substance and/or any of the excipients).
14. Patients with ataxia telangiectasia.
15. Upon the Investigator's discretion, evidence of any other medical conditions (such as psychiatric illness, physical examination or laboratory findings) that may interfere with the planned PCI treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
16. Patients planning to have or who have recently had vaccination with a live vaccine.
17. Patients concurrently receiving treatment with phenytoin.
18. Male patients unwilling to use highly effective contraception or female patients of childbearing potential unwilling to use highly effective form of contraception. Patients must continue the use of contraception during PCI treatment and subsequent chemotherapy for at least 6 months thereafter.
19. Women who are breastfeeding or who have a positive pregnancy test at baseline.
20. Patients with inadequate bone marrow function (absolute neutrophil count <1.5 x 10^9/L; platelet count <100 x 10^9/L; haemoglobin <6 mmol/L [transfusion allowed]).
21. Inadequate liver function despite satisfactory drainage (serum bilirubin persisting at >5 x upper limit of normal for the institution; aspartate aminotransferase or alanine aminotransferase >3.0 x upper limit of normal or >5 x upper limit of normal if liver metastases are present; alkaline phosphatase levels >5.0 x upper limit of normal).
22. Inadequate renal function, as determined by local practice for patients on fractionated platinum-based chemotherapy. Patients with creatinine clearance <45 mL/min (in France: <60 mL/min) must not be included.

Other protocol-defined criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PCI Biotech, Study Director — PCI Biotech
Locations (50):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Emory University Hospital, 1365C Clifton Road NE, Atlanta, Georgia
  - University of Chicago Medical Center, 5841 South Maryland Avenue, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - The Mayo Clinic Hospital - Saint Mary's Campus, 1216 Second Street Southwest, Rochester, Minnesota
  - Baylor College of Medicine, Houston, Texas
- Belgium (2):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven
- Odense Universitetshospital, Odense, Denmark
- Tampereen yliopistollinen sairaala, Syöpätautien klinikka, Tampere, Finland
- France (4):
  - Centre Hospitalier Universitaire Grenoble Alpes - Hopital Albert Michallon, Grenoble, Cedex 09
  - CHU Angers, Angers, Cedex 9
  - CHU Dupuytren, 2 Avenue Martin Luther King, Limoges
  - Institut Gustave Roussy, Département de gastro-entérologie, Villejuif
- Germany (11):
  - Klinikum rechts der Isar der Technischen Universität München, München, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Hamburg Eppendorf, I. Medizinische Klinik und Poliklinik (Gastroenterologie mit Sektionen Infektiologie und Tropenmediz), Hamburg
  - Klinikum Landshut, Landshut
  - LAKUMED Kliniken, Landshut
  - Universität Leipzig KöR, Leipzig
  - Klinikum Mannheim Universitätsklinikum gGmbH, Mannheim
  - Klinikum der Ludwig-Maximilians-Universität MünchenKlinik, München
  - Klinikum Nürnberg Nord, Medizinische Klinik 6 - (Schwerpunkte Gastroenterologie, Hepatologie, Endokrinologie), Nuremberg
- Italy (2):
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - IRCCS Saverio de Bellis, Via Turi, 27, Castellana Grotte
- Oslo Universitetssykehus HF Radiumhospitalet, Oslo, Norway
- Poland (2):
  - Zaklad Opieki Zdrowotnej MSW z Warminsko-Mazurskim Centrum Onkologii, Olsztyn, Warmian-Masurian Voivodeship
  - Med-Polonia Sp. z o.o., Poznan
- South Korea (6):
  - National Cancer Center, 323 Ilsan-ro, Ilsandong-gu, Goyang-si, Gyeonggido
  - Pusan National University Hospital, 179 Gudeok-ro, Seo-gu, Busan
  - Kyungpook National University Chilgok Hospital, 807 Hoguk-ro, Buk-gu, Daegu
  - Asan Medical Center, 88 Olympic-ro 43-gil, Songpa-gu, Seoul
  - Severance Hospital Yonsei University Health System, 50-1, Yonsei-Ro, Seodaemun-Gu, Soeul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, 222 Banpo-Daero Seocho-gu, Soeul
- Spain (6):
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Corporacio Sanitaria Parc Tauli, Sabadell
- Karolinska Universitetssjukhuset Solna, P.O Bäckencancer, Karolinska Universitetssjukhuset, Stockholm, Stockholms Ian, Sweden
- Taiwan (3):
  - Taichung Veterans General Hospital, No. 1650 Taiwan Boulevard, Sec. 4, Taichung
  - Taipei Veterans General Hospital, No. 201, Sction 2, Shi-pai Road, Taipei
  - Chang Gung Memorial Hospital, Linkou, Dept. of Medical Oncology, 5 Fuxing Street, Guishan, Taoyuan District
- Ukraine (4):
  - MNPE of Kharkiv Regional Council Regional Clinical Specialized Dispensary of Radiation Protection, Kharkiv
  - SI Institute for General and Urgent Surgery n.a. V.T. Zaitseva of NAMS of Uktraine, Kharkiv
  - SI "National Institute of Surgery and Transplantology n.a. O.O. Shalimov " of NAMS of Ukraine, Kyiv
  - Municipal Nonprofit Enterprise City Hospital #3 of Zaporizhzhia City Council, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 41 enrolled participants, all met inclusion criteria and were randomized and included in the intent-to-great (ITT) analysis set.
Period: Overall Study
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Started | 21 | 20
Completed | 0 | 0
Not Completed | 21 | 20
Not completed — Study terminated by sponsor | 9 | 11
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Death | 5 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Analysis Set
Groups:
- PCI Treatment in Conjunction With Standard of Care (SoC): Arm A: Fimaporfin-induced photochemical internalisation (PCI) of gemcitabine complemented by gemcitabine/cisplatin chemotherapy. Length of cycle is 3 weeks with PCI treatment at Day 1.
  Fimaporfin and Gemcitabine: PCI treatment consists of IV administration of Amphinex solution for injection (investigational product) at 0.22 mg/kg dose of fimaporfin, followed 4 days later by a standard dose of gemcitabine infusion (1000 mg/m²) and intraluminal laser light application. Up to 2 PCI treatments will be given.
  Gemcitabine/Cisplatin chemotherapy: Up to 8 cycles of gemcitabine/cisplatin combination chemotherapy will be administered.
- Standard of Care (SoC): Arm B: Gemcitabine/cisplatin chemotherapy. Length of cycle is 3 weeks.
  Gemcitabine/Cisplatin chemotherapy: Up to 8 cycles of gemcitabine/cisplatin combination chemotherapy will be administered.
- Total: Total of all reporting groups
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC) | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (7.30) | 64.4 (11.43) | 66.3 (9.61)
Age, Customized [Count of Participants; unit: Participants]
  <50 years of age | 0 | 2 | 2
  50 to <65 years of age | 6 | 7 | 13
  >=65 years of age | 15 | 11 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 14 | 9 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 11 | 22
  African American | 0 | 0 | 0
  Asian | 10 | 9 | 19
  Other | 0 | 0 | 0
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: From date of randomisation to date of objective disease progression or death, whichever comes first (in months)
Time Frame: Up to 18 months
Population: Modified intent-to-treat (mITT) analysis set (all randomized participants who received at least 1 dose of study treatment and had a RECIST assessment at baseline).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 19 | 15
Months | 7.29 [6.00 to 12.00] | 8.08 [6.00 to 12.00]
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); Test type: Superiority; The HR was estimated using an unstratified cox-proportional hazards model using the Efron approach for handling ties (Efron 1977), together with the associated 95% confidence intervals (CI) for the HR based on the Wald method. The effect of treatment is summarized by the hazard ratio (HR) together with its corresponding 95% Wald CI for the mITT population. No p-value will be reported

2. Secondary Outcome: Overall Survival (OS)
Description: From date of randomisation to date of death from any cause (in months)
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 19 | 15
Participants | 12 | 13
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); OS was analyzed using the modified intent-to-treat (mITT) analysis set, which included all randomized participants who received at least 1 dose of study treatment and had a RECIST assessment at baseline. Kaplan Meier Curve (KM) analysis of OS was completed for the mITT population, but the number of events was too small to draw any conclusions; Test type: Superiority; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Best Overall Response (BOR)
Description: Best response recorded from start of treatment until disease progression/recurrence (according to RECIST 1.1)
Time Frame: Up to 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 19 | 15
Participants
  Complete response | 0 | 0
  Partial response | 3 | 3
  Stable disease | 12 | 11
  Progressive disease | 4 | 1
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); BOR is summarized by randomized treatment group using the mITT analysis set; Test type: Superiority; The BOR is the best response recorded from the start of the treatment until disease progression or until the last evaluable assessment in the absence of progression. If a patient received subsequent anti-cancer therapy prior to progression, then BOR was calculated up to the point of starting the anti-cancer therapy

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Proportion of patients with measurable disease at baseline who have at least one visit response with a complete response (CR) or partial response (PR) noted (according to RECIST 1.1)
Time Frame: Up to 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 19 | 15
Participants | 3 | 3
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); Test type: Superiority; The ORR is calculated as the proportion of patients who have at least one visit response with a complete response (CR) or partial response (PR). Objective responses do not require confirmation in a randomized study. Data obtained up until progression, or last evaluable assessment in the absence of progression, will be included in the analysis of ORR. Data obtained up until progression or subsequent therapy, or last evaluable assessment in the absence of progression or subsequent therapy, will be included in the analysis of ORR

5. Secondary Outcome: Duration of Response (DoR)
Description: From first documented tumour response until first documented disease progression, or death in the absence of disease progression (in months)
Time Frame: Up to 24 months
Measure: Number; unit: Days
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 3 | 3
Days
  Patient A | 169 | NA — Patient enrolled in Arm A: PCI treatment in conjunction with Standard of Care (SoC)
  Patient B | 260 | NA — Patient enrolled in Arm A: PCI treatment in conjunction with Standard of Care (SoC)
  Patient C | 264 | NA — Patient enrolled in Arm A: PCI treatment in conjunction with Standard of Care (SoC)
  Patient D | NA — Patient enrolled in Arm B: Standard of Care (SoC) | 85
  Patient E | NA — Patient enrolled in Arm B: Standard of Care (SoC) | 1
  Patient F | NA — Patient enrolled in Arm B: Standard of Care (SoC) | 1
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); The DoR was calculated only for those with a documented response of CR or PR and is defined as the time from the date of first documented tumor response until the first date of documented disease progression or death, whichever is earlier; Test type: Superiority; DoR is listed only. In Arm A, the duration of response was 169 days in 1 participant before radiological progression was seen. In the other 2 participants in Arm A, the events were censored at 260 and 264 days, respectively. In Arm B, the duration of response was 85 days in 1 participant before radiological progression was seen. In the other 2 participants in Arm B, the events were censored at 1 day due to the early termination of the study

6. Secondary Outcome: Overall Disease Control Rate (DCR)
Description: Proportion of patients with BOR of CR, PR or stable disease (SD) (according to RECIST 1.1) at or after the first follow-up scan, partial response or complete response
Time Frame: 6 months and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 19 | 15
Participants
  Overall Disease Control Rate | 15 | 14
  Disease Control Rate at 6 Months | 11 | 10
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); DCR is reported and includes any patient with a best response of stable disease, PR or CR; Test type: Superiority; The DCR and associated exact 95% CI is summarized for the mITT population. This was repeated for DCR-6, defined as the proportion of patients with CR, PR or SD at 6 months (recorded at least 24 weeks (+/-1 week) after randomization of study treatment and prior to any PD event)

7. Secondary Outcome: Change in Tumor Size
Description: Best overall percentage change in tumour size from baseline
Time Frame: Up to 18 months
Population: Only patients with measurable disease at baseline are included in this summary.
Measure: Mean (Standard Deviation); unit: Percentage Change in Tumor Size
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 17 | 11
Percentage Change in Tumor Size | -12.06 (28.008) | -14.73 (16.377)
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); Change in tumor size in percentage was summarized for the subset of patients in the mITT analysis set who had measurable disease at baseline; Test type: Superiority; Tumor size is defined as the sum of the longest diameters (SoDs) of the RECIST 1.1 target lesions. Change in tumor size is defined as the best overall percentage change in tumor size from baseline. Percentage change in tumor size was determined for patients with measurable disease at baseline and was derived at each visit by the percentage change in the SoDs of target lesions compared to baseline

8. Secondary Outcome: Loco-regional Tumour-related Events and Biliary Complications
Description: Frequency and severity of loco-regional tumour related events and biliary complications
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 18 | 16
Participants | 12 | 8
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); Test type: Superiority; Safety, including the incidence and characteristics of biliary/loco-regional tumour-related events leading to hospitalisation and/or interventions, will be summarised descriptively

9. Secondary Outcome: Adverse Events (AEs)/Serious Adverse Events (SAEs)
Description: Number and proportion of patients with AEs/SAEs
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 18 | 16
Participants | 12 | 8
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); Test type: Superiority; Safety events leading to hospitalisation and/or interventions, will be summarised descriptively

10. Secondary Outcome: Area Under the Plasma Concentration Curve (AUC) Was Performed for Patients in Arm A.
Description: A non-compartmental analysis (NCA) was applied on the data. AUC from time zero to the last measured concentration (AUC 0-t) was initially estimated by the linear trapezoidal method.
Time Frame: Time Frame AUC calculated from time zero to C5-D8 (3 months from the first PCI treatment)
Population: AUC was calculated for each single patient and not for the population since the study was terminated and the amount of data was limited. No mean and standard deviation was calculated for the population
Measure: Number; unit: (ng/ml)*hrs
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC)
Number analyzed (Participants) | 13
(ng/ml)*hrs
  101-01 1st dose | 1017672
  101-01 2nd dose | 1399905
  101-02 | 385730
  101-03 1st dose | 576835
  101-03 2nd dose | 600546
  106-01 1st dose (No samples taken before 90 hrs, therefore AUC values is likely underestimated) | 677373
  106-01 2nd dose | 874614
  111-02 1st dose | 492274
  111-02 2nd dose | NA — One data point was measured post injection and AUC could not be calculated.
  181-06 1st dose | 566460
  181-06 2nd dose | NA — Three data points was measured post injection. Two samples were measured in the distribution phase (30 min, 4 hours) , and only one sample was measured in the elimination phase (96 hours), AUC could therefore not be calculated.
  183-03 1st dose | 751771
  183-03 2nd dose | 475001
  183-03 3rd dose | 646845
  187-02 1st dose | 709053
  187-02 2nd dose | 383882
  192-01 | 805049
  303-01 1st dose | 434347
  303-01 2nd dose | NA — The interval between the two first measured samples post injection was too long to calculate AUC. No samples were measured between 30 min and approximately 7 weeks.
  303-02 1st dose | 681663
  303-02 2nd dose | 730864
  401-01 | 521326
  501-01 | 549955

11. Secondary Outcome: Maximum Observed Concentration (Cmax) Was Performed for Patients in Arm A.
Description: A non-compartmental analysis (NCA) was applied on the data.
Time Frame: Timepoints for pharmacokinetic (PK) sampling: Day -4 (before, 30m and 4hrs after Amphinex), C1-D1, C1-D8, C2-D8, C3-D8, C4-D8, C4-D18 (before, 30m and 4hrs after Amphinex), C5-D1, and C5-D8
Population: Maximum observed concentration (Cmax) was performed for patients in arm A.
Measure: Number; unit: ng/ml
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC)
Number analyzed (Participants) | 13
ng/ml
  101-01 1st dose | 2462
  101-01 2nd dose | 2377
  101-02 | 2631
  101-03 1st dose | 2495
  101-03 2nd dose | 3172
  106-01 1st dose (No samples taken before 90 hrs, Cmax value likely underestimated) | 800
  106-01 2nd dose | 2923
  111-02 1st dose | 2221
  111-02 2nd dose | 3255
  181-06 1st dose (No sample at 30 minutes, Cmax is likely underestimated) | 1427
  181-06 2nd dose | 2321
  183-03 1st dose | 2624
  183-03 2nd dose | 2187
  183-03 3rd dose | 2571
  187-02 1st dose | 2750
  187-02 2nd dose | 1937
  192-01 | 2017
  303-01 1st dose | 2606
  303-01 2nd dose | 1848
  303-02 1st dose | 2868
  303-02 2nd dose | 3124
  401-01 | 2912
  501-01 | 2300

12. Secondary Outcome: Time to Cmax (Tmax) Was Performed for Patients in Arm A.
Description: A non-compartmental analysis (NCA) was applied on the data as described by Gabrielsson & Weiner (Methods in molecular biology, 929:161-180, 2012).
Time Frame: Timepoints for PK sampling: Day -4 (before, 30 min and 4 hours after Amphinex), C1-D1, C1-D8, C2-D8, C3-D8, C4-D8, C4-D18 (before, 30 min and 4 hours after Amphinex) , C5-D1, and C5-D8
Population: A standard non-compartmental PK analysis (NCA) of bioanalytical data from 13 patients dosed with fimaporfin was performed for the RELEASE study.
Measure: Number; unit: hours
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC)
Number analyzed (Participants) | 13
hours
  101-01 1st dose | 0.50
  101-01 2nd dose | 0.50
  101-02 | 0.50
  101-03 1st dose | 0.50
  101-03 2nd dose | 0.50
  106-01 1st dose (No samples taken before 90 hrs, erroneous data) | 90
  106-01 2nd dose | 0.50
  111-02 1st dose | 0.50
  111-02 2nd dose | 0.50
  181-06 1st dose (No sample at 30 minutes) | 4
  181-06 2nd dose | 0.50
  183-03 1st dose | 0.50
  183-03 2nd dose | 0.50
  183-03 3rd dose | 0.50
  187-02 1st dose | 0.50
  187-02 2nd dose | 0.50
  192-01 | 0.50
  303-01 1st dose | 0.50
  303-01 2nd dose | 0.50
  303-02 1st dose | 0.50
  303-02 2nd dose | 0.50
  401-01 | 0.50
  501-01 | 0.50

13. Secondary Outcome: Health-related Quality of Life (QoL)
Description: QoL assessment. Patients select one of four answers to 22 questions ranging from 1 (not at all) to 4 (very much). Lower total scores indicate a more favorable QoL perception than a higher score.
Time Frame: Up to 18 months
Population: The RELEASE study did not collect QoL data.
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: PCI Treatment in Conjunction With Standard of Care (SoC) vs Standard of Care (SoC); Test type: Superiority; As this study was terminated early, a reduced statistical analysis was conducted, and the HRQoL analyses were not conducted

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed during chemotherapy, an average of 128.3 days (range 28 to 203 days). All-Cause Mortality was monitored/assessed up to 24 months.
Description: A total of 41 participants were randomised and included in the intent-to-treat (ITT) analysis set, with 34 participants being included in the safety analysis set (18 in Arm A and 16 in Arm B) and 34 participants being included in the mITT analysis set (19 in Arm A and 15 in Arm B). The difference in the number of participants in each arm between the safety analysis set and the mITT is due to 1 participant who was randomized to Arm A but received Arm B treatment.
Arm/Group | PCI Treatment in Conjunction With Standard of Care (SoC) | Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 7/19 | 2/15
Serious Adverse Events (participants affected / at risk) | 12/18 | 8/16
Other Adverse Events (participants affected / at risk) | 18/18 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCI Treatment in Conjunction With Standard of Care (SoC) (N=18) | Standard of Care (SoC) (N=16)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 6 (9) | 3 (7)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stent malfunction (Product Issues) | 2 (4) | 1 (2)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCI Treatment in Conjunction With Standard of Care (SoC) (N=18) | Standard of Care (SoC) (N=16)
Gastrointestinal disorders (Gastrointestinal disorders) | 10 (30) | 12 (35)
General disorders and administration site conditions (General disorders) | 9 (13) | 8 (13)
Investigations (Investigations) | 6 (45) | 1 (10)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (8) | 3 (12)
Hepatobiliary disorders (Hepatobiliary disorders) | 4 (8) | 3 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8 (16) | 3 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (7) | 6 (7)
Infections and infestations (Infections and infestations) | 5 (8) | 1 (1)
Nervous system disorders (Nervous system disorders) | 6 (9) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (9) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Product issues (Product Issues) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 3 (3)
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 2 (2) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early termination of this study, no definitive conclusions can be drawn since an insufficient number of participants was recruited. A reduced statistical analysis was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04099888/Prot_SAP_000.pdf